CLINICAL TRIAL: NCT03174847
Title: Prospective Study Assessing Blood Pressure, Cardiovascular, Endothelial and Other Outcomes poSt-surgical and Medical Treatment in Patients With Primary Aldosteronism
Brief Title: Prospective Study Assessing Blood Pressure and Other Outcomes Post-treatment in Patients With Primary Aldosteronism
Acronym: PA_PACES
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PA_PACES; CHF2016.02-P (Other Grant/Funding Number: Changi Health Fund (Ltd))
Record Dates: First submitted 2017-05-26; First posted 2017-06-05 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Primary Aldosteronism; Primary Aldosteronism Due to Aldosterone Producing Adenoma; Primary Aldosteronism Due to Adrenal Hyperplasia (Bilateral)
Keywords: Primary aldosteronism; Blood pressure; Adrenalectomy; Mineralocorticoid-receptor Antagonists; Cardiovascular; Endothelial; Renal
MeSH Terms: conditions — Hyperaldosteronism | interventions — Adrenalectomy; Mineralocorticoid Receptor Antagonists; Spironolactone; Eplerenone; Amiloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples Adrenal vein blood samples (during adrenal vein sampling) Adrenal tissue (post-adrenalectomy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical Treatment: Patients who undergo medical treatment, in view of bilateral PA, or unilateral PA not keen for surgery, or indeterminate (lack of localisation on tests)
  Interventions: Drug: Mineralocorticoid Receptor Antagonists
- Surgical Treatment: Patients with unilateral PA who underwent adrenalectomy
  Interventions: Procedure: Adrenalectomy

INTERVENTIONS:
Procedure: Adrenalectomy — Adrenalectomy for unilateral adrenal hyperplasia / adenoma
  Groups: Surgical Treatment
Drug: Mineralocorticoid Receptor Antagonists — Medical treatment with MRA / amiloride
  Other Names: Spironolactone; Eplerenone; Amiloride
  Groups: Medical Treatment

SUMMARY:
Majority of patients with hypertension have primary hypertension (without an underlying cause). Secondary hypertension (due to an underlying disease) is important to recognize, as treatment can lead to cure of hypertension. Primary aldosteronism (PA) is the most common cause of secondary hypertension, and can be found in 5-10% of patients locally.

PA is caused by excessive release of a hormone (aldosterone) from the adrenal glands, which can be unilateral (one gland) or bilateral (both glands). Distinction between two is crucial as unilateral disease is treated with the aim of cure by surgery, and bilateral disease is treated by medication.

It has been shown that excess aldosterone has other harmful effects in addition to hypertension, such as directly affecting the heart, blood vessels, kidneys, diabetes and quality of life. This is supported by studies showing reversal of these effects after treatment for PA. In addition, improvements after surgery appears to be superior to medical treatment, although studies have found variable results.

Hence, the investigators aim to accurately subtype patients with PA into unilateral or bilateral disease and study the post-treatment response after both surgery and medicine with regards to the effects on blood pressure, cardiovascular, renal, metabolic and quality of life.

ELIGIBILITY:
Inclusion Criteria:

i. Legally capacitated ii. 21-80 years iii. Diagnosed with primary aldosteronism iv. Patient is willing, or has undergone, adrenal surgery (in case of unilateral disease), or medical treatment (if not keen for surgery, medically unfit, or has bilateral disease)

Exclusion Criteria:

i. Unable to give consent ii. < 21 years or > 80 years iii. Glucocorticoid remediable aldosteronism iv. Adrenal Carcinoma v. Severe or terminal medical condition(s) that in the view of the investigator prohibits participation in the study or interferes with possible treatment or health-related quality of life, e.g. cancer, end-stage liver disease, end stage renal failure vi. Female patients who are pregnant, intending to become pregnant or breastfeeding

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed primary aldosteronism
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Change from Baseline Blood Pressure at 12 months
  Blood pressure assessed by 24hr ambulatory BP

SECONDARY OUTCOMES:
Use of antihypertension medications | Change from Baseline Antihypertension medications at 12 months
  Use of antihypertension medications as expressed in daily defined dosages and total number of medications
Blood Pressure | Change from Baseline Clinic Blood Pressure at 12 months
  Clinic blood pressure
Cardiac function | Change from Baseline Cardiac function at 12 months.
  Cardiac function using 2DE
Left ventricular hypertrophy | Change from Baseline Left ventricular hypertrophy at 12 months
  as assessed by 2DE and ECG
Renal Function | Change from Baseline Renal Function at 12 months
  change in serum creatinine, calculated GFR, albuminuria (prevalence and severity)
Quality of Life (RAND-36) | Change from Baseline Quality of Life RAND-36 at 12 months
  RAND-36
Quality of Life ( Beck's depression inventory II) | Change from Baseline Quality of Life (BDI-II) at 12 months
  Beck's depression inventory II
Quality of Life (EQ5D) | Change from Baseline EQ5D at 12 months
  EQ5D
Lipids | Change from Baseline Lipids at 12 months
  Lipids
Transaminitis | Change from Baseline transaminitis at 12 months
  ALT, AST,
Insulin Resistance | Change from Baseline Insulin resistance at 12 months
  Measured with HOMA
Fasting glucose | Change from Baseline Fasting glucose at 12 months
  Fasting glucose
weight | Change from Baseline weight at 12 months
  change in weight
Control of hypertension | Change from Baseline Status of hypertension control at 12 months
  Proportion of patients reaching normal BP (ambulatory /home BP <135/85 or clinic BP <140/90)
Cure of Primary aldosteronism | Change from Baseline Status of primary aldosteronism at 12 months
  Proportion of patients with cure of PA after adrenalectomy

CONTACTS AND LOCATIONS:
Overall Officials: Troy Puar, MRCP (UK), Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Puar TH, Cheong CK, Foo RSY, Saffari SE, Tu TM, Chee MR, Zhang M, Ng KS, Wong KM, Wong A, Ng FC, Aw TC, Khoo J, Gani L, King T, Loh WJ, Soh SB, Au V, Tay TL, Tan E, Mae L, Yew J, Tan YK, Tong KL, Lee S, Chai SC. Treatment of Primary Aldosteronism and Reversal of Renin Suppression Improves Left Ventricular Systolic Function. Front Endocrinol (Lausanne). 2022 Jun 30;13:916744. doi: 10.3389/fendo.2022.916744. eCollection 2022. PMID 35846272